CLINICAL TRIAL: NCT04536012
Title: Gamification-Augmented Home-Based Exercise for Peripheral Artery Disease (GAMEPAD)
Brief Title: Gamification-Augmented Home-Based Exercise for Peripheral Artery Disease
Acronym: GAMEPAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 835034
Record Dates: First submitted 2020-08-27; First posted 2020-09-02 (Actual); Results first posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Via the Way to Health platform, all patients will receive daily text messages that inform them of their previous day's step count for 24 weeks.
- Intervention (Experimental): Participants have a 4-week ramp-up towards their step goal and are asked to maintain the goal for the rest of the study. They receive daily texts informing them if they met their step goal and biweekly texts to encourage walking for exercise.
  Participants are entered into a game. Each week they receive 70 points. If the step goal was met they keep their points. If not, they lose 10 points. At the end of the week if they have at least 40 points they move up a level. If not, they drop a level. Participants start in the middle of 5 levels.
  Participants choose a support partner who gets a weekly email with the participant's progress. We hold a 3-way phone call with the participant and partner to discuss ways they can help the participant meet their goal. Every 8 weeks, we have a follow up call if the participant is stuck in a lower level and restart them back at the middle level.
  In the follow-up period, participants continue to get a daily text stating if they met their step goal.
  Interventions: Behavioral: Gamification and Social Incentives

INTERVENTIONS:
Behavioral: Gamification and Social Incentives — Participants in the intervention arm will receive gamification and social incentives as part of the intervention. See arm descriptions for more detail.
  Arms: Intervention

SUMMARY:
A randomized trial of a gamification-enhanced home-based walking program compared with a standard home-based walking program in patients with intermittent claudication. Patients will be provided with a Fitbit device and set an exercise goal. Over the next 16 weeks, patients will receive text message reminders to exercise and daily steps will be tracked. Half of patients will be randomized to a gamified interface that leverages behavioral economic principles to encourage exercise.

DETAILED DESCRIPTION:
Peripheral artery disease, atherosclerotic vascular disease involving the lower extremities, leads to functional limitation by causing leg pain with ambulation (intermittent claudication). Supervised exercise programs improve walking endurance in patients with intermittent claudication, but many patients are unable to travel to centers for treatment. In a recent trial, a home-based exercise program using wearable fitness trackers and telephone coaching failed to increase walking distance in patients with intermittent claudication, but this intervention did not leverage gamification or health behavior theory. Therefore, a randomized controlled trial was proposed comparing a gamification-enhanced home-based walking program with an attention control in patients with intermittent claudication. Patients in both arms will be provided with a wearable fitness tracker, wear the tracker for 2 weeks to establish a baseline daily step count and set a goal for step increase by the end of the 16-week study period. Patients in the attention control arm will receive daily text messages with a report of their previous day's step count. Patients in the gamification intervention arm will receive automated coaching via daily text messages and the intervention will also involve a precommittment pledge, slow ramp-up of step goals, weekly progression (or regression) through levels with loss-framing of points, and support from a family member or friend. After 16 weeks, change in daily step counts from baseline will be compared between study arms. Secondary behavioral phenotyping analyses will be undertaken to identify psychometric features associated with response to the gamification intervention.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Peripheral artery disease, defined as ankle-brachial index < 0.90, lower extremity CT scan or ultrasound consistent with PAD, angiography with ≥ 70% stenosis in any lower extremity artery, or a history of medical or surgical revascularization
* Owns a smartphone or tablet operating the iOS or Android operating system

Exclusion Criteria:

* Unable or unwilling to provide informed consent, including but not limited to cognitive or language barriers (reading or comprehension)
* Critical limb ischemia, defined as rest pain, ulceration, or tissue loss involving the lower extremity
* Planned lower extremity revascularization
* Prior above or below the knee amputation
* Require a wheelchair or the use of a walking aid other than a cane
* Currently participating in a supervised exercise program for patients with PAD
* Anticipated life expectancy less than 6 months
* Any other reason why it is not feasible to complete the entire 6-month study
* Step count > 7500/day during the baseline data collection period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2024-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Fanaroff, MD, MHS, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fanaroff AC, Coratti S, Farraday D, Norton L, Rareshide C, Zhu J, Levin MG, Damrauer SM, Giri JS, Chokshi NP, Jackson BM, Patel MS. Effect of Gamification Plus Automated Coaching to Increase Physical Activity Among Patients With Peripheral Artery Disease: The GAMEPAD Randomized Controlled Trial. J Am Heart Assoc. 2025 Dec 16;14(24):e038921. doi: 10.1161/JAHA.124.038921. Epub 2025 Dec 3. PMID 41334739
- [Derived] Fanaroff AC, Coratti S, Farraday D, Norton L, Rareshide C, Zhu J, Levin MG, Damrauer SM, Giri JS, Chokshi NP, Jackson BM, Patel MS. Gamification-augmented home-based exercise for peripheral artery disease: Rationale and design of the GAMEPAD Study. Am Heart J. 2024 Apr;270:95-102. doi: 10.1016/j.ahj.2024.02.003. Epub 2024 Feb 13. PMID 38354997

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Participants have a 4-week ramp-up towards their step goal and are asked to maintain the goal for the rest of the study. They receive daily texts informing them if they met their step goal and biweekly texts to encourage walking for exercise.
  Participants are entered into a game. Each week they receive 70 points. If the step goal was met they keep their points. If not, they lose 10 points. At the end of the week if they have at least 40 points they move up a level. If not, they drop a level. Participants start in the middle of 5 levels.
  Participants choose a support partner who gets a weekly email with the participant's progress. We hold a 3-way phone call with the participant and partner to discuss ways they can help the participant meet their goal. Every 8 weeks, we have a follow up call if the participant is stuck in a lower level and restart them back at the middle level.
  In the follow-up period, participants continue to get a daily text stating if they met their step goal.
  Gamification and Social Incentives: Participants in the intervention arm will receive gamification and social incentives as part of the intervention. See arm descriptions for more detail.
Period: Overall Study
Arm/Group | Control | Intervention
Started | 52 | 51
Completed | 51 | 45
Not Completed | 1 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 52 | 51 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (9.1) | 69.4 (8.2) | 69.7 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 22 | 49
  Male | 25 | 29 | 54
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 42 | 39 | 81
  Black | 6 | 10 | 16
  Asian | 2 | 0 | 2
  Hispanic | 0 | 1 | 1
  Other | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 52 | 51 | 103
Education [Count of Participants; unit: Participants]
  Some high school | 2 | 0 | 2
  High school graduate | 7 | 7 | 14
  Some college | 11 | 22 | 33
  College graduate | 32 | 22 | 54
Education [Count of Participants; unit: Participants]
  Some High School | 2 | 0 | 2
  High School Graduate | 7 | 7 | 14
  Some College | 11 | 22 | 33
  College Graduate | 32 | 22 | 54
Marital Status [Count of Participants; unit: Participants]
  Single | 8 | 11 | 19
  Married | 27 | 30 | 57
  Other | 17 | 10 | 27
Annual Household Income [Count of Participants; unit: Participants]
  < $50,000 | 17 | 18 | 35
  $50,000 to $100,000 | 19 | 15 | 34
  > $100,000 | 16 | 18 | 34
Prior Use of Smartphone or Wearable to Track Steps [Count of Participants; unit: Participants] | 35 | 27 | 62
Current Smoking [Count of Participants; unit: Participants] | 7 | 4 | 11
Hypertension [Count of Participants; unit: Participants] | 37 | 46 | 83
Hyperlipidemia [Count of Participants; unit: Participants] | 37 | 36 | 73
Diabetes [Count of Participants; unit: Participants] | 17 | 20 | 37
Prior MI [Count of Participants; unit: Participants] | 16 | 10 | 26
Stroke [Count of Participants; unit: Participants] | 8 | 4 | 12
Heart Failure [Count of Participants; unit: Participants] | 7 | 5 | 12
COPD [Count of Participants; unit: Participants] | 7 | 12 | 19
Kidney Disease [Count of Participants; unit: Participants] | 10 | 10 | 20
San Diego Claudication Questionnaire [Count of Participants; unit: Participants]
  Classic Claudication | 9 | 12 | 21
  Atypical Leg Pain | 26 | 27 | 53
  No Symptoms | 17 | 12 | 29
Baseline Daily Step Count [Mean (Standard Deviation); unit: Steps] | 4540 (2379) | 4191 (1627) | 4367 (2039)
Goal Step Increase [Mean (Standard Deviation); unit: Steps] | 1160 (2033) | 1549 (740) | 1353 (1541)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.4 (7.2) | 30.8 (5.4) | 30.1 (6.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Daily Step Count
Description: Change in daily step count from baseline to the intervention period (main adjusted model)
Time Frame: 16 Weeks
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | Control | Intervention
Number analyzed (Participants) | 52 | 51
steps per day | 783 (2441) | 1770 (2481)

2. Secondary Outcome: Change in Daily Step Count
Description: Change in daily step count from baseline to the follow-up period (main adjusted model)
Time Frame: 24 Weeks
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | Control | Intervention
Number analyzed (Participants) | 52 | 51
steps per day | 717 (2410) | 1786 (2476)

3. Other Pre Specified Outcome: Change in Walking Impairment Questionnaire Score
Description: Change in Walking Impairment Questionnaire score from baseline to the end of the intervention period, and from baseline to the end of the follow-up period.
  Participants are asked to rate the degree of difficulty of various physical activities, ranging from 0 (unable) to 4 (no difficulty). Scores are divided by the maximum number of points and presented on a scale of 0%-100% where 0% indicates they are unable to do the activity and 100% indicates they have no difficulty.
Time Frame: 24 Weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 52 | 51
units on a scale
  WIQ Distance | -3.8 [-12.2 to 4.5] | 7.3 [-1.5 to 16]
  WIQ Speed | 1.7 [-5 to 8.5] | 4.8 [-2.3 to 11.8]
  WIQ Stair Climbing | 6.4 [-1 to 13.8] | 9.5 [1.8 to 17.2]
  WIQ Overall | 1.4 [-5 to 7.8] | 5.7 [-3.5 to 15]

4. Other Pre Specified Outcome: Change in PROMIS Mobility, Pain Interference, and Satisfaction With Social Roles and Activities Scores
Description: Change in PROMIS (Patient-Reported Outcomes Measurement Information System) mobility, pain interference, and satisfaction with social roles and activities scores from baseline to the end of the intervention period, and from baseline to the end of the follow-up period.
  In the mobility survey, participants are asked to rate the level of difficulty of various physical activities on a scale from 1 to 5, where 1 means they are unable to do the activity and 5 means they have no difficulty. In the pain interference survey, they are asked to rate the degree to which pain interfered with various activities on a scale from 1 to 5, where 1 indicates pain did not interfere and 5 indicates pain very much interfered. For the satisfaction with social roles, participants are asked to rate how satisfied they are with their ability to perform various activities on a scale of 1-5, where 1 indicates they are not satisfied and 5 indicates they are very satisfied.
Time Frame: 24 Weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 52 | 51
units on a scale
  PROMIS Pain | -2.2 [-4.5 to 0.2] | -4.7 [-7.2 to -2.3]
  PROMIS Social Function | -0.6 [-2.8 to 1.6] | 0.3 [-2 to 2.6]

5. Other Pre Specified Outcome: Change in SF-36 Physical Functioning Scale
Description: Change in SF-36 (36-Item Short Form Survey) physical functioning scale from baseline to the end of the intervention period, and from baseline to the end of the follow-up period. Participants are asked to self-report their health using 8 variously scaled scores. The scales are re-coded to values from 0 to 100, with 0 indicating lowest functioning/well-being and 100 indicating the highest.
Time Frame: 24 Weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 52 | 51
units on a scale
  Physical functioning | 0.3 [-4.4 to 5] | 6.7 [1.8 to 11.6]
  Role functioning/physical | 5.9 [-3.9 to 15.6] | 12.8 [2.6 to 23]
  Role functioning/emotional | 5.7 [-6.2 to 17.6] | 3.9 [-8.5 to 16.3]
  Energy/fatigue | 3 [-1.4 to 7.4] | 3 [-1.6 to 7.7]
  Emotional well-being | 0.9 [-3.3 to 5] | 2.4 [-1.9 to 6.7]
  Social functioning | 7.4 [-0.5 to 15.4] | 2 [-6.3 to 10.4]
  Pain | 3.5 [-2.2 to 9.2] | 10.5 [4.5 to 16.4]
  General Health | 1.2 [-2.5 to 4.8] | 4.2 [0.4 to 8]
  Health Change | 5.3 [-2.4 to 13] | 16.9 [8.8 to 24.9]

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: Adverse events were collected via participant reports through study surveys at 16 weeks, and 24-weeks or participant reports to study staff through text, email or phone call.
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/52 | 1/51
Serious Adverse Events (participants affected / at risk) | 3/52 | 6/51
Other Adverse Events (participants affected / at risk) | 13/52 | 21/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=52) | Intervention (N=51)
Orthopedic (Musculoskeletal and connective tissue disorders) | 0 | 5
Cardiovascular (Cardiac disorders) | 1 | 1
Fitbit-related (Product Issues) | 0 | 0
Other (General disorders) | 2 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=52) | Intervention (N=51)
Orthopedic (Musculoskeletal and connective tissue disorders) | 5 | 8
Cardiovascular (Cardiac disorders) | 1 | 4
Fitbit-related (Product Issues) | 3 | 0
Other (General disorders) | 8 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/12/NCT04536012/Prot_SAP_000.pdf